CLINICAL TRIAL: NCT05822128
Title: Sleepiness in the Elderly: Validation of the Alternative Epworth Sleepiness Scale ESS-ALT in French
Brief Title: Alternative Epworth Sleepiness Scale ESS-ALT in French
Acronym: SOMNOLD
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230377
Record Dates: First submitted 2023-03-27; First posted 2023-04-20 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Excessive Daytime Sleepiness
Keywords: Excessive daytime sleepiness; Elderly; Epworth Sleepiness Scale
MeSH Terms: conditions — Disorders of Excessive Somnolence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Seniors with suspected sleep disorders referred for assessment: Seniors with suspected sleep disorders referred for assessment
  Interventions: Other: Test of an alternative Epworth Sleepiness Scale ESS-ALT in French

INTERVENTIONS:
Other: Test of an alternative Epworth Sleepiness Scale ESS-ALT in French — Seniors recruited into the study will test the Epworth Alternate Sleepiness Scale -ALT

SUMMARY:
The Epworth Sleepiness Scale (ESS) is undoubtedly the most commonly used tool in daily clinical practice to assess daytime sleepiness in patients of all ages by means of a self-administered questionnaire.

In elderly subjects, the clinician is often confronted with difficulties in accurately estimating the ESS score and measuring subjective daytime sleepiness. Indeed, according to Onen et al, the ESS tends to underestimate the prevalence of sleep disorders in the geriatric population, mainly due to non-response to problematic items, namely:

* Item 3: Sitting, inactive in a public place (cinema, theater, meeting)
* Item 8: In a car that has been stopped for a few minutes.

In order to overcome this problem, Janine Gronewold's German team has developed and begun work on the validation of an alternative version of the ESS, the ESS-ALT, adapted to the population of interest, in German.

The aim of the present work is to adapt the ESS-ALT in French, then to study its correlation with sleep data recorded by nocturnal polysomnography, and among the secondary objectives, to correlate it with sleep latency during iterative sleep latency tests, in order to propose to the clinician a simple, reproducible tool, allowing to measure daytime sleepiness in elderly subjects.

DETAILED DESCRIPTION:
Developed in 1991 by Dr. Johns at the University of Melbourne and modified by him in 1997, the Epworth Sleepiness Scale (ESS) is undoubtedly the most commonly used tool in daily clinical practice to assess daytime sleepiness in patients of all ages by means of a self-administered questionnaire.

In elderly subjects, the clinician is often confronted with difficulties in accurately estimating the ESS score and measuring subjective daytime sleepiness. Indeed, according to Onen et al, the ESS tends to underestimate the prevalence of sleep disorders in the geriatric population, mainly due to non-response to problematic items, namely:

* Item 3: Sitting, inactive in a public place (cinema, theater, meeting)
* Item 8: In a car that has been stopped for a few minutes.

In order to overcome this problem, Janine Gronewold's German team has developed and begun work on the validation of an alternative version of the ESS, the ESS-ALT, adapted to the population of interest, in German.

The aim of the present work is to adapt the ESS-ALT in French, then to study its correlation with sleep data recorded by nocturnal polysomnography, and among the secondary objectives, to correlate it with sleep latency during iterative sleep latency tests, in order to propose to the clinician a simple, reproducible tool, allowing to measure daytime sleepiness in elderly subjects

ELIGIBILITY:
Inclusion Criteria:

* Patient 65 years of age and older
* Consulting for sleep disorders
* Enrolled in a social security system or entitled to it
* Patient informed and having expressed his non-opposition to participate in the research

Exclusion Criteria:

* Severe psychiatric or cognitive disorders that do not allow the completion of examinations/questionnaires
* Patients who are dependent for all acts of daily life
* Patients with a very short life expectancy
* Patients under guardianship or curatorship
* Patients under AME
* Patients whose first language is not French
* Patients with visual or cognitive impairments that make reading impossible

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Seniors with suspected sleep disorders referred for assessment
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Validation of the alternative Epworth Daytime Sleepiness Scale -ALT adapted to the elderly and geriatric population in French | 24 hours
  forward and backward translation" between English and French, and correlation with the ESS sleepiness scale.

SECONDARY OUTCOMES:
Study of the correlation between the results of the French ESS-ALT and polysomnography data | 24 hours
  Statistical comparison to identify the intrinsic validity of the ESS-ALT
Study of the correlation between the results of the French ESS-ALT and MSLT (Multiple Sleep Latency Test) data | 24 hours
  Statistical comparison to identify the intrinsic validity of the ESS-ALT
intrinsic validity of the ESS-ALT in French | 24 months
  Statistical comparison to identify the intrinsic validity of the ESS-ALT
Study of the correlation between the ESS-ALT cohort in French and the ESS-ALT cohort in Germany | 24 months
  Statistical comparison to identify the intrinsic validity of the French version of ESS-ALT

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospital Charles Foix, Ivry-sur-Seine
  - service des pathologies du sommeil, hôpital Pitié Salpêtrière, Paris